CLINICAL TRIAL: NCT01536262
Title: A Randomised, Double-blind, Parallel-group Study to Assess the Safety and Efficacy of 52 Weeks of Once Daily Treatment of Orally Inhaled Tiotropium + Olodaterol Fixed-dose Combination (2.5µg / 5µg, 5µg / 5µg ) and Olodaterol (5 µg) Delivered by the RESPIMAT Inhaler in Japanese Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Japan Long-term Safety for Tiotropium Plus Olodaterol
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1237.22
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Results first posted 2015-07-15 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — tiotropium-olodaterol; olodaterol

ARMS (3):
- Tiotropium + Olodaterol (high dose) (Other): Tiotropium and Olodaterol FDC solution for inhalation - RESPIMAT
  Interventions: Drug: Tiotropium + Olodaterol; Device: Respimat
- Olodaterol (Other): Olodaterol solution for inhalation - RESPIMAT
  Interventions: Drug: Olodaterol; Device: Respimat
- Tiotropium + Olodaterol (low dose) (Other): Tiotropium and Olodaterol FDC solution for inhalation - RESPIMAT
  Interventions: Drug: Tiotropium + Olodaterol; Device: Respimat

INTERVENTIONS:
Drug: Tiotropium + Olodaterol — Tiotropium and Olodaterol FDC once daily inhalation
  Arms: Tiotropium + Olodaterol (low dose)
Device: Respimat — Respimat inhaler
  Arms: Tiotropium + Olodaterol (low dose)
Drug: Tiotropium + Olodaterol — Tiotropium and Olodaterol FDC once daily inhalation
  Arms: Tiotropium + Olodaterol (high dose)
Drug: Olodaterol — Olodaterol once daily inhalation
  Arms: Olodaterol
Device: Respimat — Respimat inhaler
  Arms: Tiotropium + Olodaterol (high dose)
Device: Respimat — Respimat inhaler
  Arms: Olodaterol

SUMMARY:
The primary objective of this study is to assess the safety of 52 weeks once daily treatment with orally inhaled tiotropium + olodaterol FDC and olodaterol (delivered by the RESPIMAT Inhaler) in Japanese patients with Chronic Obstructive Pulmonary Disease (COPD).

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of chronic obstructive pulmonary disease.
2. Relatively stable airway obstruction with post FEV1< 80% predicted normal and post FEV1/FVC <70%.
3. Male or female Japanese patients, 40 years of age or older.
4. Smoking history of more than 10 pack years.

Exclusion criteria:

1. Significant disease other than COPD
2. Clinically relevant abnormal lab values.
3. History of asthma.
4. Diagnosis of thyrotoxicosis
5. Diagnosis of paroxysmal tachycardia
6. History of myocardial infarction within 1 year of screening visit
7. Unstable or life-threatening cardiac arrhythmia.
8. Hospitalization for heart failure within the past year.
9. Known active tuberculosis.
10. Malignancy for which patient has undergone resection, radiation therapy or chemotherapy within last five years
11. History of life-threatening pulmonary obstruction.
12. History of cystic fibrosis.
13. Clinically evident bronchiectasis.
14. History of significant alcohol or drug abuse.
15. Thoracotomy with pulmonary resection
16. Oral ß-adrenergics.
17. Oral corticosteroid medication at unstable doses
18. Regular use of daytime oxygen therapy for more than one hour per day
19. Pulmonary rehabilitation program in the six weeks prior to the screening visit
20. Investigational drug within one month or six half lives (whichever is greater) prior to screening visit
21. Known hypersensitivity to ß-adrenergic drugs, anticholinergics, BAC, EDTA
22. Pregnant or nursing women.
23. Women of childbearing potential not using a highly effective method of birth control
24. Patients who are unable to comply with pulmonary medication restrictions
25. Patients with narrow-angle glaucoma or micturition disorder due to prostatic hyperplasia etc.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2012-02; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (24):
- Japan (24):
  - 1237.22.81015 Boehringer Ingelheim Investigational Site, Chiyoda-ku, Tokyo
  - 1237.22.81023 Boehringer Ingelheim Investigational Site, Chuo-ku, Tokyo
  - 1237.22.81009 Boehringer Ingelheim Investigational Site, Hamamatu, Shizuoka
  - 1237.22.81011 Boehringer Ingelheim Investigational Site, Kishiwada, Osaka
  - 1237.22.81007 Boehringer Ingelheim Investigational Site, Komatsu, Ishikawa
  - 1237.22.81028 Boehringer Ingelheim Investigational Site, Koriyama, Fukushima
  - 1237.22.81019 Boehringer Ingelheim Investigational Site, Koto-ku,Tokyo
  - 1237.22.81021 Boehringer Ingelheim Investigational Site, Kyoto, Kyoto
  - 1237.22.81014 Boehringer Ingelheim Investigational Site, Minami-ku, Kumamoto, Kumamoto
  - 1237.22.81017 Boehringer Ingelheim Investigational Site, Morioka, Iwate
  - 1237.22.81004 Boehringer Ingelheim Investigational Site, Nagaoka, Niigata
  - 1237.22.81029 Boehringer Ingelheim Investigational Site, Nagasaki, Nagasaki
  - 1237.22.81027 Boehringer Ingelheim Investigational Site, Osakasayama, Osaka
  - 1237.22.81008 Boehringer Ingelheim Investigational Site, Saku, Nagano-ken
  - 1237.22.81001 Boehringer Ingelheim Investigational Site, Sapporo, Hokkaido
  - 1237.22.81016 Boehringer Ingelheim Investigational Site, Sapporo, Hokkaido
  - 1237.22.81022 Boehringer Ingelheim Investigational Site, Sapporo, Hokkaido
  - 1237.22.81025 Boehringer Ingelheim Investigational Site, Sapporo, Hokkaido
  - 1237.22.81018 Boehringer Ingelheim Investigational Site, Setagaya-ku, Tokyo
  - 1237.22.81026 Boehringer Ingelheim Investigational Site, Tagajyo,Miyagi
  - 1237.22.81010 Boehringer Ingelheim Investigational Site, Takatsuki, Osaka
  - 1237.22.81020 Boehringer Ingelheim Investigational Site, Toyohashi, Aichi
  - 1237.22.81030 Boehringer Ingelheim Investigational Site, Unzen, Nagasaki
  - 1237.22.81003 Boehringer Ingelheim Investigational Site, Yokohama,Kanagawa

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was a 52-week multi-centre, randomised, double-blind and parallel-group design.
Groups:
- Olodaterol (5 μg): Olodaterol solution for inhalation - RESPIMAT: 2 Oral inhalation once daily in the morning up to 52-week treatment period.
- Tiotropium + Olodaterol (2.5 / 5 μg): Tiotropium and Olodaterol fixed dose combination (FDC) solution for inhalation - RESPIMAT : 2 Oral inhalation once daily in the morning up to 52-week treatment period.
- Tiotropium + Olodaterol (5 / 5 μg): Tiotropium and Olodaterol fixed dose combination (FDC) solution for inhalation - RESPIMAT: 2 Oral inhalation once daily in the morning up to 52-week treatment period.
Period: Overall Study
Arm/Group | Olodaterol (5 μg) | Tiotropium + Olodaterol (2.5 / 5 μg) | Tiotropium + Olodaterol (5 / 5 μg)
Started | 41 | 40 | 41
Completed | 33 | 38 | 39
Not Completed | 8 | 2 | 2
Not completed — Adverse Event | 6 | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — Other than stated above | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): This patient set included all patients who received at least 1 dose of treatment.
Groups:
- Tiotropium + Olodaterol (2.5 / 5 μg); Tiotropium + Olodaterol (5 / 5 μg): Tiotropium and Olodaterol FDC solution for inhalation - RESPIMAT : 2 Oral inhalation once daily in the morning up to 52-week treatment period.
- Total: Total of all reporting groups
Arm/Group | Olodaterol (5 μg) | Tiotropium + Olodaterol (2.5 / 5 μg) | Tiotropium + Olodaterol (5 / 5 μg) | Total
Number analyzed (Participants) | 41 | 40 | 41 | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.5 (7.2) | 70.0 (7.5) | 68.1 (7.1) | 69.9 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 3 | 5
  Male | 40 | 39 | 38 | 117

OUTCOME MEASURES:

1. Primary Outcome: Number (%) of Patients With Drug-related AEs
Description: Number (%) of patients with drug-related Adverse Events (AEs).
Time Frame: From first drug administration until 21 days after the last administration, upto 392 days
Population: Treated set: This patient set included all patients who received at least 1 dose of treatment.
Measure: Number; unit: percentage of participants
Groups:
- Tiotropium + Olodaterol (5 / 5 μg): Tiotropium and Olodaterol FDC solution for inhalation - RESPIMAT: 2 Oral inhalation once daily in the morning up to 52-week treatment period.
Arm/Group | Olodaterol (5 μg) | Tiotropium + Olodaterol (2.5 / 5 μg) | Tiotropium + Olodaterol (5 / 5 μg)
Number analyzed (Participants) | 41 | 40 | 41
percentage of participants | 4.9 | 5.0 | 7.3

2. Secondary Outcome: FEV1 AUC0-3h Response
Description: Forced Expiratory Volume in 1 second Area Under Curve (AUC0-3h) response. FEV1 AUC0-3h was calculated using the trapezoidal rule, divided by the duration (3 h) to report in litres. Baseline was defined as the mean of the 2 pre-treatment FEV1 values measured on day 1 (-1 hour and -10 minutes) prior to administration of the first dose of study drug.
  Note: The Mean presented is the unadjusted mean.
Time Frame: Baseline and 1 h, 10 min pre-dose and 30 min, 1 h, 2 h, 3 h post-dose after 52 weeks
Population: Full analysis set (FAS): This patient set included all randomised patients who received at least 1 dose of treatment and had both non-missing baseline and at least 1 non-missing post-baseline efficacy measurement. Assignment to FAS was done after implementation of any data handling rules which set measurements to missing.
Measure: Mean (Standard Error); unit: L
Arm/Group | Olodaterol (5 μg) | Tiotropium + Olodaterol (2.5 / 5 μg) | Tiotropium + Olodaterol (5 / 5 μg)
Number analyzed (Participants) | 34 | 39 | 39
L | 0.132 (0.030) | 0.260 (0.031) | 0.237 (0.024)

3. Secondary Outcome: Trough FEV1 Response
Description: Trough Forced Expiratory Volume in 1 second Response. The trough was defined as the mean of the 1 h pre-dose and 10 min pre-dose measurements after 52 weeks. Baseline was defined as the mean of the 2 pre-treatment FEV1 values measured on day 1 (-1 hour and -10 minutes) prior to administration of the first dose of study drug.
  Note: The Mean presented is the unadjusted mean.
Time Frame: Baseline and 1 h, 10 min pre-dose after 52 weeks
Population: Full analysis set (FAS)
Measure: Mean (Standard Error); unit: L
Arm/Group | Olodaterol (5 μg) | Tiotropium + Olodaterol (2.5 / 5 μg) | Tiotropium + Olodaterol (5 / 5 μg)
Number analyzed (Participants) | 34 | 39 | 39
L | 0.075 (0.027) | 0.168 (0.031) | 0.143 (0.025)

ADVERSE EVENTS:
Time Frame: From first drug administration until 21 days after the last administration, upto 392 days.
Arm/Group | Olodaterol (5 μg) | Tiotropium + Olodaterol (2.5 / 5 μg) | Tiotropium + Olodaterol (5 / 5 μg)
Serious Adverse Events (participants affected / at risk) | 5/41 | 6/40 | 3/41
Other Adverse Events (participants affected / at risk) | 21/41 | 20/40 | 24/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Olodaterol (5 μg) (N=41) | Tiotropium + Olodaterol (2.5 / 5 μg) (N=40) | Tiotropium + Olodaterol (5 / 5 μg) (N=41)
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Olodaterol (5 μg) (N=41) | Tiotropium + Olodaterol (2.5 / 5 μg) (N=40) | Tiotropium + Olodaterol (5 / 5 μg) (N=41)
Constipation (Gastrointestinal disorders) | 3 | 1 | 4
Bronchitis (Infections and infestations) | 3 | 5 | 6
Nasopharyngitis (Infections and infestations) | 17 | 11 | 11
Pharyngitis (Infections and infestations) | 1 | 3 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.